CLINICAL TRIAL: NCT00051324
Title: Neurobiological Predictors of Huntington's Disease Trial
Brief Title: Neurobiological Predictors of Huntington's Disease (PREDICT-HD)
Acronym: PREDICT-HD
Status: Active, not recruiting | Type: Observational
Sponsor: Jordan Schultz (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Jordan Schultz, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 199904075; R01NS040068 (NIH)
Record Dates: First submitted 2003-01-08; First posted 2003-01-09 (Estimated); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Huntington Disease
Keywords: Huntington's disease; Huntington disease; HD
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebral spinal fluid acquired and retained since 2012.
  Urine, plasma and cell lines to be acquired and retained since study initiation 2002.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this trial is to study early brain and behavioral changes in people who have the gene expansion for Huntington's disease, but are currently healthy and have no symptoms.

DETAILED DESCRIPTION:
Huntington's Disease (HD) is an inherited disease that causes changes in a person's ability to control movements, thinking, and feelings. The intent of this study is to learn more about the beginning changes in thinking skills, emotional regulation, and brain structure and function as a person begins the transition from health to HD.

Preliminary studies indicate that people with HD may have marked decline before an actual diagnosis. This study will help reveal the earliest indicators of the disease and what factors influence the age at which a person carrying the gene develops the disease. It is necessary to get information on the early stages of HD in order to develop drugs that can slow or postpone the onset of HD. The investigators hope this study will provide essential information for future trials of experimental drugs for HD.

During this study, participants will undergo several detailed tests, including MRI scans of the brain, cognitive assessments, physical exams, bio specimen (blood, urine, cerebral spinal fluid) collection and neurological and psychiatric testing.

ELIGIBILITY:
Inclusion Criteria:

* men and women at risk for HD, who have been tested for the HD gene mutation, and who have not been diagnosed with symptoms of HD (CAG ≥36 for CAG-expanded group or CAG <36 for CAG-norm group).

Exclusion Criteria:

* diagnosis of manifest HD (at least 50% confidence by neurologist that symptoms are present);
* clinical evidence of unstable medical or psychiatric illness (including substance abuse);
* history of sever learning disability or mental retardation;
* history of other CNS disease or event (e.g., seizures or head trauma);
* current treatment with antipsychotic medications, including the traditional neuroleptics such as haloperidol as well as the atypical antipsychotics risperidone, clozapine, quetiapine, and olanzapine;
* treatment with phenothiazine-derivative antiemetic medications such as prochlorperazine, metoclopramide, promethazine, and Inapsine on a regular basis (greater than 3 times per month);

Specific exclusion criteria for the lumbar puncture:

* Current use of anti-coagulants
* Current use of anti-platelets
* Unable to provide consent for him/herself

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People at risk for HD, who have been tested for the HD gene mutation, and who have not been diagnosed with symptoms of HD.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2002-08; Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Refine the prediction of disease diagnosis (motor conversion) | One year
  HD diagnosis will be better predicted by adding longitudinal change to the baseline measures of striatal and white matter volumes, tone-paced and speeded tapping score, stroop interference and motor score.
Characterize disease progression prior to diagnosis. | One year
  Document change scores for each marker using its slope.
  Comparisons of change rates across time will suggest measures best suited to clinical trials by large effect sizes and low variability.
Establish possible validity and reliability of disease measures. | One year
  This will require that we continuously analyze recently collected data, remove items that are insensitive, and add new items to be tested throughout the course of the study. The power and sensitivity of future multi-site trials and studies depend on accurate measures of marker validity.
  HD diagnosis will be better predicted by UHDRS total motor score following new standardized reliability training and by the tapping task under modified more challenging, conditions. Psychiatric and functional ratings will be improved with item response analyses and dynamic piloting of item edits to establish the most psychometrically sound items for clinical trials.

OTHER OUTCOMES:
Cerebral spinal fluid containing unique biomarker signatures. | One year
  Lumbar puncture is conducted at the University of Iowa
Cerebral spinal fluid biomarker changes correlating with HD progression. | One year
  Lumbar puncture is conducted at the University of Iowa

CONTACTS AND LOCATIONS:
Overall Officials: Jane S. Paulsen, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All data have been de-identified and anonymized with the best possible methods to allow and facilitate data sharing with other investigators. Data has been shared to CHDI and dbGaP.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be on dbGaP and at CHDI for data sharing with no anticipated endpoint.
Access Criteria: NINDS monitors dbGaP and CHDI scientific staff monitors their data copy.

REFERENCES:
- [Derived] Chelsky D, Joyce C, Bockholt HJ, Rudnick PA, Adams WH, McAllister F, Smock JW, Newton MA, Paulsen JS. Discovery and Targeted Proteomic Studies Reveal Striatal Markers Validated for Huntington's Disease. Ann Clin Transl Neurol. 2025 Dec 9. doi: 10.1002/acn3.70272. Online ahead of print. PMID 41363816
- [Derived] Paulsen JS, Lourens S, Kieburtz K, Zhang Y. Sample enrichment for clinical trials to show delay of onset in huntington disease. Mov Disord. 2019 Feb;34(2):274-280. doi: 10.1002/mds.27595. Epub 2019 Jan 14. PMID 30644132
- [Derived] Reed ER, Latourelle JC, Bockholt JH, Bregu J, Smock J, Paulsen JS, Myers RH; PREDICT-HD CSF ancillary study investigators. MicroRNAs in CSF as prodromal biomarkers for Huntington disease in the PREDICT-HD study. Neurology. 2018 Jan 23;90(4):e264-e272. doi: 10.1212/WNL.0000000000004844. Epub 2017 Dec 27. PMID 29282329
- [Derived] Epping EA, Kim JI, Craufurd D, Brashers-Krug TM, Anderson KE, McCusker E, Luther J, Long JD, Paulsen JS; PREDICT-HD Investigators and Coordinators of the Huntington Study Group. Longitudinal Psychiatric Symptoms in Prodromal Huntington's Disease: A Decade of Data. Am J Psychiatry. 2016 Feb 1;173(2):184-92. doi: 10.1176/appi.ajp.2015.14121551. Epub 2015 Oct 16. PMID 26472629
- See also: PREDICT-HD YouTube Channel — http://www.youtube.com/user/PREDICTHD